CLINICAL TRIAL: NCT06377787
Title: Effects of ELDOA in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01732 Aneeqa Zaheer
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cervicogenic Headache
Keywords: ELDOA; Cervicogenic Headache; Cervical spine
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA and conventional therapy (Experimental): hot pack and TENS for10 min, cervical PIR (MET) in flexion, extension, side bending and rotation (single set of 4rep with 6 sec hold once a day) and ELDOA method C0-C1-C2, C2 & C3 positions for cervical spine (2 sets of five repetitions with 45 sec hold and 15sec rest between each set once a day).
  Interventions: Other: ELDOA and conventional therapy
- conventional therapy (Other): hot pack and TENS for 10 minutes, cervical PIR (MET) in flexion, extension, side bending and rotation (single set of 4 reps with 6 seconds hold once a day).
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: ELDOA and conventional therapy — hot pack and TENS for10 min, cervical PIR (MET) in flexion, extension, side bending and rotation (single set of 4rep with 6 sec hold once a day) and ELDOA method C0-C1-C2, C2 & C3 positions for cervical spine (2 sets of five repetitions with 45 sec hold and 15sec rest between each set once a day).
  Arms: ELDOA and conventional therapy
Other: conventional therapy — include hot pack and TENS for 10 minutes, cervical PIR (MET) in flexion, extension, side bending and rotation (single set of 4 reps with 6 seconds hold once a day).
  Arms: conventional therapy

SUMMARY:
The aim of our study is to determine the effect of ELDOA in relieving pain, improving ROM and functional disability in patients with cervicogenic headache. This study will add to the growing body of knowledge that if this technique yields comparable outcomes, it would be the alternative therapy. Moreover, it would add to the society as no literature is available on the effect of ELDOA technique in the management of Cervicogenic headache.

DETAILED DESCRIPTION:
Cervicogenic Headache (CEH) is mainly caused by neck or paravertebral soft tissue lesions. It is chronic headache that arises from the Atlanto-occipital and upper cervical joints and is perceived in one or more regions of the head or face. One of the known treatment options that create decompression at spinal segment level is called ELDOA it is described as a conditioning method involving a series of movements and body stretches to help correct body posture, rehabilitate people with injuries and prevent injuries

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-45 years
* Both male and female.
* Onset of pain > 4 weeks.
* Flexion rotation test positive with estimated rotation range reduced by more than 10 degrees from the anticipated normal range (44 degrees)
* Tenderness of upper three cervical joints.
* Presence of active trigger points in upper trapezius and sub occipital extensors.

Exclusion Criteria:

* Hypertension.
* Recent (<6 months) whiplash injury and other cervical soft tissue injuries.
* History of cervical spinal vertebrae fracture.
* Positive sharp purser test
* Acute disc protrusion • History of cancer.
* Previous surgical intervention of head, neck and thoracic spine

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
(Numeric Pain Rating Scale). | four weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable while the NPRS exhibited moderate reliability (ICC = 0.27-0.84)
NDI (U) (Neck Disability Index) | four weeks
  The neck disability index is a ten-item self-reported questionnaire that assesses pain and associated disability, with a total max score of 50 points . An Urdu version of neck disability index will use in this study. An intra-class correlation coefficient (ICC) revealed excellent test-retest reliability for all items (ICC = 0.86-0.98) and total scores (ICC = 0.99) of the NDI-U.
Inclinometer | four weeks
  Cervical range of motion will be measured using inclinometer. It is a common instrument used to measure joint range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University; Asghar Khan, Study Chair — Riphah International University
Locations (1):
- Alkhidmat Raazi Hospital CBR Town, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No